CLINICAL TRIAL: NCT00002863
Title: PHASE I FEASIBILITY TRIAL OF CRYOSURGICAL ABLATION OF SOFT TISSUE SARCOMAS OF THE EXTREMETY
Brief Title: Cryosurgery in Treating Patients With Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065134; LAC-USC-11S-96-1; NCI-V96-1059
Record Dates: First submitted 1999-11-01; First posted 2004-07-07 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Sarcoma
Keywords: recurrent childhood rhabdomyosarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; previously untreated childhood rhabdomyosarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Drug Therapy; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chemotherapy
Procedure: conventional surgery
Procedure: cryosurgery

SUMMARY:
RATIONALE: Cryosurgery kills cancer cells by freezing them. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining cryosurgery with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of cryosurgery with or without chemotherapy in treating patients who have soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the safety and morbidity associated with cryosurgical ablation in patients with soft tissue sarcomas of the extremity.

OUTLINE: All patients undergo 1 session of cryoablation. Patients with high-grade sarcoma receive systemic chemotherapy 10-14 days after cryoablation at the discretion of the consulting medical oncologist, and undergo surgery 2-3 weeks following chemotherapy. Patients with low-grade sarcoma and those with high-grade sarcoma who do not receive chemotherapy undergo surgery 4-6 weeks after cryoablation. Surgery for all patients consists of en bloc resection or amputation, with limb salvage attempted when feasible. Patients are followed weekly for 3 weeks.

PROJECTED ACCRUAL: A total of 12 patients (approximately 6 patients with low-grade, high-risk sarcoma and 6 with high-grade sarcoma) will be entered over approximately 6 months. The study will be suspended for the following: vascular complication that requires surgical intervention for correction in 2 patients; any neuropraxia that shows no evidence of resolution after 3 months in 2 patients; any wound complication that requires surgical correction in 4 patients; or any deep wound infection that requires surgical drainage in 4 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven soft tissue sarcoma (STS) of the extremity Review by Pathology Department of the University of Southern California CT or MRI required prior to biopsy Disease in one of the following categories: High-grade tumor Low-grade tumor at high risk for local recurrence, i.e.: Adjacent to bone or vital neurovascular structures and able to be removed with a minimal surgical margin (i.e., plane of dissection goes through reactive zone of tumor) Lesion more than 5 cm in diameter The following tumors exclude: Primary sarcoma of the bone Metastatic carcinoma STS of the head and neck Visceral STS, e.g., breast, uterus, spermatic cord, mediastinum chest wall STS of the pelvis or retroperitoneum

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Hematopoietic: WBC at least 3,000 Platelets at least 75,000 Hemoglobin at least 9 g/Dl Hepatic: Bilirubin no greater than 1.5 mg/dL AST/ALT no greater than 2.5 times normal Renal: Not specified Other: No concurrent disease that renders patient medically or psychologically unable to tolerate treatment

PRIOR CONCURRENT THERAPY: At least 30 days since therapy for sarcoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1996-06; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Menendez, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States